CLINICAL TRIAL: NCT04060563
Title: Frequency Specific Microcurrent for the Treatment of Diastasis Recti
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment too slow.
Sponsor: Diana Trang (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Diana Trang, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20190124H
Record Dates: First submitted 2019-08-13; First posted 2019-08-19 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Diastasis Recti
Keywords: diastasis recti; postpartum; family medicine; microcurrent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham (fake) microcurrent therapy (Sham Comparator): Sham (fake) microcurrent therapy (placing the microcurrent pads on the patient and turning the microcurrent box on placebo mode )
  Interventions: Device: INSPIRSTAR IS02 MICROCURRENT STIMULATOR
- Frequency specific microcurrent therapy (Experimental): Frequency specific microcurrent therapy (100-300μA microccurrent amps) with Diastasis Recti Repair protocol (8),
  Interventions: Device: INSPIRSTAR IS02 MICROCURRENT STIMULATOR

INTERVENTIONS:
Device: INSPIRSTAR IS02 MICROCURRENT STIMULATOR — Investigators will use the Inspirstar microcurrent stimulator TENS device. It is an FDA 510k approved portable hand-held device used for the symptomatic relief of chronic pain. It generates low current intensity pulses in the ranges of 20μA to 400μA.
  For this study, investigators will use a treatment range of 100-300μA. Frequency specific microcurrent therapy (100-300μA microccurrent amps) with Diastasis Recti Repair protocol (8), times 2 treatments for a consistent total of 11 hours 32 minutes.

SUMMARY:
Determine if frequency specific microcurrent therapy improves pain management of DRA by 30% or greater.

DETAILED DESCRIPTION:
Females aged 18 years or older who are postpartum from a singleton gestation status post vaginal and with diastasis recti will be recruited. The aim of this study is to determine if frequency specific microcurrent therapy improves pain management of DRA by 30% or greater

Improving DRA after microcurrent therapy in post-partum females may allow a faster, more effective return to activity thereby improving the return-to-duty transition and establishing personal readiness by meeting military fitness standards.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Active Duty and DoD beneficiary Postpartum Females (12 hours to 24 hours) with Diastasis Rectus Abdominus (DRA) pain
* Aged 18 years or older
* Singleton gestation/delivered (one baby carried and born)
* Vaginal delivery
* Nulliparous (first pregnancy) or multiparous (more than one pregnancy in the past)

Exclusion Criteria:

* less than 18 years of age
* females greater than 24 hours post-partum
* Medical history to include pacemaker
* History of arrhythmia
* Transplant status
* Insulin pump
* Pain pump
* Active cancer
* Inability to measure IRD
* Delivery via caesarean section
* Operative vaginal delivery (vacuum or forceps)
* 3rd or 4th degree vaginal laceration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data

REFERENCES:
- [Background] Benjamin DR, van de Water AT, Peiris CL. Effects of exercise on diastasis of the rectus abdominis muscle in the antenatal and postnatal periods: a systematic review. Physiotherapy. 2014 Mar;100(1):1-8. doi: 10.1016/j.physio.2013.08.005. Epub 2013 Oct 5. PMID 24268942
- [Background] Chiarello CM, McAuley JA, Hartigan EH. Immediate Effect of Active Abdominal Contraction on Inter-recti Distance. J Orthop Sports Phys Ther. 2016 Mar;46(3):177-83. doi: 10.2519/jospt.2016.6102. Epub 2016 Jan 26. PMID 26813756
- [Background] Fernandes da Mota PG, Pascoal AG, Carita AI, Bo K. Prevalence and risk factors of diastasis recti abdominis from late pregnancy to 6 months postpartum, and relationship with lumbo-pelvic pain. Man Ther. 2015 Feb;20(1):200-5. doi: 10.1016/j.math.2014.09.002. Epub 2014 Sep 19. PMID 25282439
- [Background] Keshwani N, Mathur S, McLean L. Validity of Inter-rectus Distance Measurement in Postpartum Women Using Extended Field-of-View Ultrasound Imaging Techniques. J Orthop Sports Phys Ther. 2015 Oct;45(10):808-13. doi: 10.2519/jospt.2015.6143. Epub 2015 Aug 24. PMID 26304645
- [Background] Keshwani N, Mathur S, McLean L. Relationship Between Interrectus Distance and Symptom Severity in Women With Diastasis Recti Abdominis in the Early Postpartum Period. Phys Ther. 2018 Mar 1;98(3):182-190. doi: 10.1093/ptj/pzx117. PMID 29228344
- [Background] Liaw LJ, Hsu MJ, Liao CF, Liu MF, Hsu AT. The relationships between inter-recti distance measured by ultrasound imaging and abdominal muscle function in postpartum women: a 6-month follow-up study. J Orthop Sports Phys Ther. 2011 Jun;41(6):435-43. doi: 10.2519/jospt.2011.3507. Epub 2011 Feb 2. PMID 21289454
- [Background] Sancho MF, Pascoal AG, Mota P, Bo K. Abdominal exercises affect inter-rectus distance in postpartum women: a two-dimensional ultrasound study. Physiotherapy. 2015 Sep;101(3):286-91. doi: 10.1016/j.physio.2015.04.004. Epub 2015 May 6. PMID 26094117
- [Background] Goossen, S., Demitry, P. (2018) Frequencies for Physical Therapy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated early at 13/160 subjects enrolled due to slow enrollment. 1 subject screenfailed.
Groups:
- Sham (Fake) Microcurrent Therapy: Sham (fake) microcurrent therapy (placing the microcurrent pads on the patient and turning the microcurrent box on placebo mode )
  INSPIRSTAR IS02 MICROCURRENT STIMULATOR: Investigators will use the Inspirstar microcurrent stimulator TENS device. It is an FDA 510k approved portable hand-held device used for the symptomatic relief of chronic pain. It generates low current intensity pulses in the ranges of 20μA to 400μA.
  For this study, investigators will use a treatment range of 100-300μA. Frequency specific microcurrent therapy (100-300μA microccurrent amps) with Diastasis Recti Repair protocol (8), times 2 treatments for a consistent total of 11 hours 32 minutes.
- Frequency Specific Microcurrent Therapy: Frequency specific microcurrent therapy (100-300μA microccurrent amps) with Diastasis Recti Repair protocol (8),
  INSPIRSTAR IS02 MICROCURRENT STIMULATOR: Investigators will use the Inspirstar microcurrent stimulator TENS device. It is an FDA 510k approved portable hand-held device used for the symptomatic relief of chronic pain. It generates low current intensity pulses in the ranges of 20μA to 400μA.
  For this study, investigators will use a treatment range of 100-300μA. Frequency specific microcurrent therapy (100-300μA microccurrent amps) with Diastasis Recti Repair protocol (8), times 2 treatments for a consistent total of 11 hours 32 minutes.
Period: Overall Study
Arm/Group | Sham (Fake) Microcurrent Therapy | Frequency Specific Microcurrent Therapy
Started | 4 | 8
Completed | 3 | 6
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: No analysis was conducted due to study termination for slow enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham (Fake) Microcurrent Therapy | Frequency Specific Microcurrent Therapy | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 5 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Inter-rectus Distances (IRD)
Description: Investigator will apply ultrasound gel and measure Inter-rectus distances (IRD) -- via ultrasound or if unable via ultrasound, via palpation and measuring tape -- taken at 4 locations using the medial margins of both rectus abdominis muscles:
  A. 2.5 cm above the umbilical ring, B. upper margin of the umbilical ring, C. lower margin of the umbilical ring, and D. 2.5 cm below the umbilical ring.
  A and D were recorded.
Time Frame: screening (pre and post initial treatment)
Population: No subject data was analyzed by a biostatistician due to study termination for slow/lack of enrollment. Raw data are reported.
Measure: Mean (Full Range); unit: centimeters
Arm/Group | Sham (Fake) Microcurrent Therapy | Frequency Specific Microcurrent Therapy
Number analyzed (Participants) | 4 | 8
centimeters
  inter-rectus distance 2.5 cm above umbilical ring (pre) | 4.74 [3.89 to 6.83] | 3.88 [2.71 to 4.97]
  inter-rectus distance 2.5 cm above umbilical ring (post) | 4.89 [3.64 to 7.62] | 3.3 [1.91 to 4.45]
  inter-rectus distance 2.5 cm below umbilical ring (pre) | 2.23 [1.16 to 3.49] | 1.85 [1.25 to 2.62]
  inter-rectus distance 2.5 cm below umbilical ring (post) | 2.14 [1.13 to 3.07] | 1.84 [1.06 to 2.05]

2. Primary Outcome: Inter-rectus Distances (IRD)
Description: as for outcome 1
Time Frame: visit 2/week 2
Population: No subject data was analyzed by a biostatistician due to study termination for slow/lack of enrollment. Raw data are reported. 1 sham subject was lost to followup.
Measure: Mean (Full Range); unit: centimeters
Arm/Group | Sham (Fake) Microcurrent Therapy | Frequency Specific Microcurrent Therapy
Number analyzed (Participants) | 4 | 8
centimeters
  inter-rectus distance 2.5 cm above umbilical ring: number analyzed (Participants) | 3 | 8
  inter-rectus distance 2.5 cm above umbilical ring | 3.42 [3.17 to 3.66] | 2.46 [.93 to 3.79]
  inter-rectus distance 2.5 cm below umbilical ring: number analyzed (Participants) | 3 | 8
  inter-rectus distance 2.5 cm below umbilical ring | 1.46 [0.89 to 1.89] | 1.68 [0.71 to 4.25]

3. Primary Outcome: Inter-rectus Distances (IRD)
Description: as for outcome 1
Time Frame: visit 3/week 3
Population: No subject data was analyzed by a biostatistician due to study termination for slow/lack of enrollment. Raw data are reported. 1 sham subject lost to followup. 2 intervention subjects lost to followup.
Measure: Mean (Full Range); unit: centimeters
Arm/Group | Sham (Fake) Microcurrent Therapy | Frequency Specific Microcurrent Therapy
Number analyzed (Participants) | 4 | 8
centimeters
  inter-rectus distance 2.5 cm above umbilical ring: number analyzed (Participants) | 3 | 6
  inter-rectus distance 2.5 cm above umbilical ring | 3.1 [2.23 to 3.46] | 2.16 [1.25 to 3.76]
  inter-rectus distance 2.5 cm below umbilical ring: number analyzed (Participants) | 3 | 6
  inter-rectus distance 2.5 cm below umbilical ring | 1.28 [0.79 to 1.86] | 1.56 [0.33 to 3.76]

ADVERSE EVENTS:
Time Frame: Duration of subject participation: 12 weeks.
Arm/Group | Sham (Fake) Microcurrent Therapy | Frequency Specific Microcurrent Therapy
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 0/4 | 0/8

LIMITATIONS AND CAVEATS:
This study was terminated due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT04060563/Prot_SAP_002.pdf